# STATISTICAL ANALYSIS PLAN: INDV-6000-405

**Protocol Title:** A Single-Dose Study to Evaluate the Relative Bioavailability, Safety, and Tolerability of SUBLOCADE at Alternative Injection Locations in Adults

Final Version: 23 Oct 2023

**NCT:** NCT05704543

# STATISTICAL ANALYSIS PLAN Title Page

Protocol Title: A Single-Dose Study to Evaluate the Relative Bioavailability, Safety, and

Tolerability of SUBLOCADE at Alternative Injection Locations in Adults

Protocol Number: INDV-6000-405

Product: SUBLOCADE® (buprenorphine extended-release) injection

Short Title: SUBLOCADE Alternative Injection Locations

Sponsor Name: Indivior Inc.

Legal Registered Address: Indivior Inc., 10710 Midlothian Turnpike, Suite 125, North

Chesterfield, VA 23235 USA

Regulatory Agency Identifier Number(s)

Registry ID: NCT05704543

Registry Name: clinicaltrial.gov

Version: 2.0

**Confidentiality Statement** 

The information contained in this document is privileged and confidential. Do not copy, circulate or otherwise distribute without written authorization from Indivior Inc.

Statistical Analysis Plan Approval

# **Table of Contents**

| LIS | T OF | TABLES | | 4 |
|---|---|---|---|---|
| LIS | T OF I | FIGURE: | S | 4 |
| 1 | INTR | ODUCT | ION | 5 |
| | 1.1 | Versio | n History | 5 |
| | 1.2 | - | tives and Endpoints | |
| | 1.3 | | Design | |
| 2 | STAT | | L HYPOTHESES | _ |
| | 2.1 | - | olicity Adjustment | |
| 3 | | | E DETERMINATION | |
| 4 | | | NS FOR ANALYSIS | |
| 5 | | | L ANALYSES | |
| | 5.1 | | al Considerations | |
| | | 5.1.1 | Timing of Analyses | |
| | | 5.1.2 | Populations for Analyses | |
| | 5.2 | | pant Dispositions | |
| | 5.3 | | ry Endpoint(s) Analysis | |
| | | 5.3.1 | Definition of endpoint(s) | |
| | | 5.3.2 | Main analytical approach | |
| | 5.4 | | dary Endpoint(s) Analysis | |
| | 5.5 | | ry/Exploratory Endpoint(s) Analysis | |
| | 5.6 | Other | Safety Analyses | |
| | | 5.6.1 | Extent of Exposure | |
| | | 5.6.2 | Adverse Events | 13 |
| | | 5.6.3 | Additional safety assessments | 14 |
| | 5.7 | Other | Analyses | 16 |
| | | 5.7.1 | Major Protocol Deviations | 16 |
| | | 5.7.2 | Demographic and Baseline Disease Characteristics | 16 |
| | | 5.7.3 | Medical and Psychiatric History | 16 |
| | | 5.7.4 | Urine Drug Screen Results | 17 |
| | | 5.7.5 | Prior and Concomitant Therapies and Medications | |
| | | 5.7.6 | Subgroup analyses | |
| | 5.8 | | n Analyses | |
| | ٠.٠ | | , | / |

| 6 | SUP | SUPPORTING DOCUMENTATION1 | |
|---|---|---|---|
| | 6.1 | Appendix 1: List of Abbreviations | |
| | 6.2 | Appendix 2: Changes to Protocol-Planned Analyses | 18 |
| | 6.3 | Appendix 3: Definition and Use of Visit Windows in Reporting | |
| | 6.4 | Appendix 4: Endpoint Derivations | |
| | | 6.4.1 PK Parameters | 18 |
| | | 6.4.2 Handling of BLQ and abberant plasma concentrations | 18 |
| | | 6.4.3 Injection site Reactions Customised MedDRA Queries (CMQ) | 19 |
| | 6.5 | Appendix 5: Methods to Manage Missing Data | 20 |
| | | 6.5.1 Adverse event data | 20 |
| | | 6.5.2 Missing Date Information for Concomitant Medications | 21 |
| | 6.6 | Appendix 6: Methods to Manage Character Values of Clinical Laboratory Pa | arameters22 |
| | 6.7 | Appendix 7: Data Set Descriptions | 22 |
| | 6.8 | Appendix 8: Concomitant Medication Definition | 23 |
| 7 | REFE | RENCES | 23 |
| | | SAP Version History Summary | |
| | | Objectives, Endpoints and Estimands | |
| | | Populations for Analysis | |
| | | Primary PK parameters | |
| | | Additional PK Parameters of BUP Following SUBLOCADE Injection | |
| | | PK Parameters of Norbuprenorphine Following SUBLOCADE Injection | |
| | | Laboratory Assessments | |
| | | List of Abbreviations | |
| | | CMQ List of Preferred Terms for Injection Site Reactions | |
| | | Definition of Prior and Concomitant Medications for Run-In Period | |
| Ta | ble 11 | Definition of Concomitant Medications for Post Injection Period | 23 |
| | | LIST OF TABLES | |
| <b>-:</b> - | | LIST OF FIGURES | • |
| FIB | ure 1 | . Study schematic | 8 |

#### 1 INTRODUCTION

SUBLOCADE is currently approved for SC administration in 4 different quadrants of the abdomen. Injection locations are rotated to minimize irritation.

Having one or more alternate injection sites is desirable in this patient population who may be taking SUBLOCADE for extended durations, based upon clinical response.

Data cited from literature suggests that the proposed alternative injection locations for SC administration are viable options for delivering similar PK properties: back of upper arm, buttocks, and thigh. Therefore, this study will assess the relative bioavailability of buprenorphine (BUP) when SUBLOCADE is administered to these alternate injection sites compared to the currently approved injection location, abdomen in participants with OUD.

#### 1.1 Version History

This Statistical Analysis Plan (SAP) for study INDV-6000-405 is based on the protocol dated 18 Nov. 2022 and eCRF dated 6 Dec. 2022. SAP approval history is shown in Table 1.

This SAP provides the detailed methodology for summary and statistical analyses of the data collected in Study INDV-6000-405. This document may modify the plans outlined in the protocol; however, any major modifications of the primary endpoint definition or its analysis will also be reflected in a protocol amendment.

**Table 1. SAP Version History Summary** 

| SAP Version | Associated Protocol Amendment | Approval Date | Change | Rationale |
|---|---|---|---|---|
| 1.0 | Not Applicable | 23OCT2023 | Not Applicable | Original version |
| 2.0 | Not Applicable | | Changed definition of prior and concomitant medication Added Appendix 8 to illustrate this definition. | To be consistent with the other studies in the portfolio. |

#### 1.2 Objectives and Endpoints

Objectives, endpoints and estimands are detailed in Table 2.

**Table 2 Objectives, Endpoints and Estimands** 

| Objective | Statistical | | | |
|---|---|---|---|---|
| Clinical Category | Category | Estimand | | |
| | | Endpoint | Population | population-level summary |
| | | pavailability of buprenorphine (BUP) when administered at a attention at single SC injection of SUBLOCADE in partic | ·- | |
| Pharmacokinetic | Primary | AUC <sub>0-28 Days</sub> of BUP plasma concentration | PK evaluable | Geometric mean ratios with 90% confidence intervals (CIs) |
| | Primary | C <sub>max</sub> of BUP plasma concentration | PK evaluable | Geometric mean ratios with 90% Cls |
| Secondary Objective: 1 | o evaluate the safet | and tolerability of SUBLOCADE when administered at altern | ative injection loc | ations, in comparison to the abdomen |
| AEs | Secondary | Proportion of participants with treatment-emergent adverse events (TEAEs) | Safety | Categorical descriptive |
| | Secondary | Proportion of participants with TEAEs identified as injection site reactions | Safety | Categorical descriptive |
| | Secondary | Proportion of participants with treatment-emergent serious adverse events (SAEs) | Safety | Categorical descriptive |
| Injection site<br>assessments | Secondary | Injection site grading at 10 minutes and 2 hours post SUBLOCADE dosing | Safety | Numeric or categorical descriptive |
| | Secondary | Injection Site Pain VAS at 1, 5, 10, 15 and 30 minutes post SUBLOCADE dosing | Safety | Numeric descriptive |

- To assess other PK parameters of BUP when administered at alternative injection locations (test treatments), in comparison to the abdomen (reference treatment) following a single SC injection of SUBLOCADE in participants with OUD
- To assess the relative bioavailability of norbuprenorphine and other norbuprenorphine PK parameters following the single SC injection of SUBLOCADE.

| Pharmacokinetic | Exploratory | AUC <sub>last</sub> of BUP plasma concentration | PK evaluable | Geometric mean ratios with 90% Cls |
|---|---|---|---|---|
| | Exploratory | T <sub>max</sub> of BUP plasma concentration | PK evaluable | Medians, ranges, descriptive |
| | Exploratory | C <sub>trough</sub> of BUP plasma concentration | PK evaluable | Numeric, descriptive |
| | Exploratory | AUC <sub>0-28 Days</sub> of norbuprenophine plasma concentration | PK evaluable | Geometric mean ratios with 90% Cls |
| | Exploratory | C <sub>max</sub> of norbuprenophine plasma concentrationfrom | PK evaluable | Geometric mean ratios with 90% Cls |
| | Exploratory | AUC <sub>last</sub> of norbuprenophine plasma concentration | PK evaluable | Geometric mean ratios with 90% Cls |
| | Exploratory | T <sub>max</sub> of norbuprenophine plasma concentration | PK evaluable | Medians, ranges, descriptive |
| | Exploratory | C <sub>trough</sub> of norbuprenophine plasma concentration | PK evaluable | Numeric, descriptive |

#### 1.3 Study Design

This is a multi-centre, randomized, open-label, single-dose, parallel-group pharmacokinetic study in participants with moderate or severe OUD (based on criteria from the DSM-5).

Participants will provide written informed consent before any protocol-related procedures commence. The study includes both a Residential (Inpatient) Period and a Non-Residential (Outpatient) Period.

Following Screening, all eligible participants must be stabilized on 12 mg SUBOXONE® (BUP/naloxone) sublingual film QD for a minimum of 7 days before the SUBLOCADE injection. Dose induction/stabilization onto SUBOXONE film may be completed as outpatient or inpatient, as necessary, according to the prescribing information.

All participants will be admitted to the residential facility by the evening of Day -3.

Following the residential period (Day -3 to Day -1), on Day 1, eligible participants will be randomized to receive a single, SC injection of 300 mg SUBLOCADE at a different injection location ie, abdomen (reference) or one of the alternative injection locations (test) ie, back of upper arm, buttocks, and thigh.

On Day -2, a blood sample will be collected prior to the SUBOXONE dose. On Day -1, blood samples will be collected prior to the SUBOXONE dose, and at 0.5, 1, 2, 4, 6, 12 hours post dose. On Day 1, blood samples will be collected prior to injection of SUBLOCADE, and at 1, 2, 4, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48 hours post dose. Blood samples will also be collected on Days 4, 6, 8, 11, 15, 18, 22, 25 and 29, as close to the time of SUBLOCADE injection performed on Day 1 as possible.

It is important that participants do not use any BUP-containing products, either therapeutically or illicitly since their use would compromise the PK assessment of BUP and its metabolite, norbuprenorphine.

Approximately 80 participants in the United States will be randomized in total, ideally to achieve 15 completed participants per each of the 4 treatment arms (injection locations): Abdomen (reference), back of upper arm, buttocks, and thigh. The total duration of the study for each participant, including Screening (up to 30 days), Treatment (up to 11 days in the Residential Period and up to 25 days in the Non-residential Period), and Follow up, will be up to approximately 66 days.

The study schematic is illustrated in Figure 1 below.

Figure 1. Study schematic



#### 2 STATISTICAL HYPOTHESES

No formal statistical hypotheses will be tested in this study. Relative bioavailability of BUP when administered to alternative injection sites (back of upper arm, buttocks, and thigh) compared to that when administered to the abdomen will be informally evaluated.

# 2.1 Multiplicity Adjustment

Not applicable, as there will be no formal hypothesis testing.

#### 3 SAMPLE SIZE DETERMINATION

No formal statistical power analysis was performed to determine the sample size of this study. Based on historical experience from previous similar clinical trials, approximately 80 randomized participants was considered adequate to achieve at least 15 PK evaluable participants per injection site location to assess the relative bioavailability of SUBLOCADE

300 mg at each of the alternate injection site locations compared to the the abdomen (the reference injection location).

#### 4 POPULATIONS FOR ANALYSIS

Data for all participants will be assessed to determine if participants meet the criteria for inclusion in each analysis population prior to releasing the database. Classifications will be documented per standard operating procedures.

The analysis populations are defined as shown in Table 3. below.

Table 3. Populations for Analysis

| Population | Description |
|---|---|
| Screened | All participants who sign the ICF. |
| Enrolled | All screened participants who receive at least 1 dose of SUBOXONE film during run-in. |
| Randomised | All enrolled participants who are randomised to one of the 4 treatment arms (injection locations). |
| PK Evaluable<br>Analysis Set | All randomised participants who receive SUBLOCADE injection and provide an adequate number of post randomization PK samples to derive key PK parameters for SUBLOCADE (ie, C <sub>max</sub> and AUC <sub>0-28 Days</sub> ). The participants will be analysed corresponding to the actual injection location used. |
| Safety Analysis Set | All enrolled participants who received SUBLOCADE injection. The participants will be analysed corresponding to the actual injection location used. |
| Run-In Safety<br>Analysis Set | All enrolled participants who receive at least 1 dose of SUBOXONE film during run-in, and same as the enrolled population |

# **5 STATISTICAL ANALYSES**

#### 5.1 General Considerations

AUC and  $C_{max}$  values will be summarized using descriptive statistics such as the geometric mean and coefficient of variation (CV%).  $T_{max}$  values will be summarized as the median, minimum, and maximum. Other continuous variables will be summarised using descriptive statistics such as mean, standard deviations (SD) and/or CV%, median, minimum, and maximum. Categorical variables will be reported as frequency counts (including number missing) and the percentage of participants in corresponding categories.

PK parameters will be derived by noncompartmental analysis with Phoenix<sup>™</sup> WinNonlin<sup>®</sup> software (Version 8.3.4 or higher, Certara, LP)<sup>1</sup> in conjunction with Certara Integral (Version 22.10.1 or higher, Certara, USA, Inc.)<sup>2</sup> using actual sampling times. SAS<sup>®</sup> software (SAS Institute, Cary, North Carolina)<sup>3</sup> will be used for the statistical analyses and the production of TFLs.

BUP and norbuprenophine plasma concentrations following SUBLOCADE injection will be summarised at each scheduled time point by injection location. The PK profile of each analyte will be summarized graphically by injection site, using both linear and semi-log plots.

Additionally, BUP and norbuprenophine plasma concentrations during the run-in period with SUBOXONE film will also be be summarised at each scheduled time point, and graphically displayed using both linear and semi-log plots.

Spaghetti plots (each individual participant's plasma concentration shown on the same plot, separate plots for each injection site location) will also be generated for both analytes. These plots will include each participant's plasma concentrations during both the inpatient portion of the run-in period and the randomized period. (ie. X-axis will range from Day -2 to Day 29).

#### **5.1.1** Timing of Analyses

Final data analysis will be performed after all BUP and norbuprenorphine PK parameters have been derived, participants belonging to each analysis population (Table 3.) documented and the database locked.

# 5.1.2 Populations for Analyses

By-timepoint summaries and graphical displays of PK profiles (e.g., buprenorphine plasma concentration) following the SUBLOCADE dose will use the Safety Analysis Set.

PK parameters following the SUBLOCADE dose will be summarized and analysed using the PK evaluable set.

All safety data (eg. TEAEs, injection site grading) following the SUBLOCADE dose will be summarized using the Safety Analysis Set.

By-timepoint summaries and graphical displays of PK profiles (e.g., buprenorphine plasma concentration) during the run-in period will use the Enrolled participant set.

All safety data during the run-in period will be summarized using the Run-In Safety Analysis Set (same as the Enrolled participant set).

#### 5.2 Participant Dispositions

The number and percentage of participants who were screened, enrolled (i.e., received at least 1 dose of SUBOXONE film), randomised and not randomised (including the reason for not randomising), will be summarized by study site and overall, using the number of participants in the screened population as the denominator.

The number and percentage of participants who received SUBLOCADE dose and completed the study, and the number and percentage of participants who belong to the PK Evaluable Set and the safety analysis set (i.e., received SUBLOCADE dose), as well as participants who discontinued early and reason, will be summarized by randomised injection site location and overall, using the number of participants in the randomised population as the denominator. If actual treatment (injection site location) received is different from the randomised treatment for any participant, dispositions will be repeated by the actual injection site location.

# 5.3 Primary Endpoint(s) Analysis

#### 5.3.1 Definition of endpoint(s)

The primary PK parameters of BUP following SUBLOCADE injection will be derived as shown in Table 4.

**Table 4. Primary PK parameters** 

| Parameter | Description |
|---|---|
| AUC <sub>0-28 Days</sub> | Area under the BUP plasma concentration-time curve from time zero (Day 1) to 28 days post-dose (Day 29), calculated by the linear trapezoidal method. |
| C <sub>max</sub> | Maximum observed plasma concentration of BUP |

#### 5.3.2 Main analytical approach

Estimand strategy: Principal stratum strategy will be used, such that only subjects with an adequate amount of PK data will be included in the analysis.

Analysis set: PK Evaluable Set

Analysis methodology: Natural log-transformed BUP  $AUC_{0-28\,Days}$  and  $C_{max}$  from SUBLOCADE Phase will be analyzed using an analysis of variance (ANOVA) model with injection site location as the independent variable. The 90% confidence interval will be estimated for the ratio of population geometric means (test/reference) corresponding to exponentiated differences in least square means.

The comparisons of interest are the three alternative injection sites (test) versus abdomen (reference; [namely: back of upper arm vs abdomen, buttocks vs abdomen, and thigh vs abdomen])

Intercurrent events and missing data: Missing values will be retained as missing in the analysis.

#### 5.4 Secondary Endpoint(s) Analysis

All secondary endpoints (i.e., safety endpoints) will be based on the Safety Analysis Set. All summaries will be by the actual injection site location and for overall. The difference to

abdomen injection location (with 95% confidence interval) will be estimated for injection locations of upper arm, buttocks, and thigh.

The following secondary endpoints will be derived as the proportion of participants reporting at least one of the specified events, and summarized using frequency counts and percentages:

- Proportion of participants with TEAEs
- Proportion of participants with TEAEs identified as injection site reactions
- Proportion of participants with treatment-emergent SAEs

TEAEs identified as injection site reactions will be summarised using customised MedDRA queries (CMQ). See Section 6.4 for the complete list of PTs for the CMQ.

Further details on Safety Analysis are detailed in Section 5.6.2.

Each component of the Injection site grading (pain, tenderness and erythema/redness, induration, swelling) at 10 minutes and 2 hours post SUBLOCADE dosing will be summarized using frequency counts and percentages of participants reporting the specific level of severity, including none (Grade 0), mild (Grade 1), moderate (Grade 2), severe (Grade 3), or potentially life threatening (Grade 4) as continuous score (0 to 4). The assessments will be tabulated according to nominal time points, with/without excluding the assessments at time points out of the assessment windows (Protocol 10.6 Appendix 6 Table 11).

Injection Site Pain Visual Analog Scale (VAS) at 1, 5, 10, 15 and 30 minutes post SUBLOCADE dosing will be summarized using descriptive statistics. The assessments will be tabulated according to nominal time points, with/without excluding the assessments at time points out of the assessment windows.

#### 5.5 Tertiary/Exploratory Endpoint(s) Analysis

The following PK parameters for SUBLOCADE will be derived as shown in Table 5. for BUP and Table 6. for norbuprenorphine. The plasma terminal half-life and AUC extrapolated to infinity  $(AUC_{0-inf})$  are not calculated as the duration of the PK evaluation is shorter than the plasma terminal half-life reported for SUBLOCADE (43-60 days).

Table 5. Additional PK Parameters of BUP Following SUBLOCADE Injection

| Parameter | Description |
|---|---|
| AUC <sub>last</sub> | Area under the BUP plasma concentration-time curve from time 0 (Day 1) to the last quantifiable BUP concentration, calculated by the linear trapezoidal method |
| T <sub>max</sub> | Time to attain the maximum observed BUP plasma concentration |
| C <sub>trough</sub> | BUP plasma concentration measured on Day 29 |

Table 6. PK Parameters of Norbuprenorphine Following SUBLOCADE Injection

| Parameter | Description |
|---|---|
| AUC <sub>0-28 Days</sub> | Area under the norbuprenorphine plasma concentration-time curve from time zero (Day 1) to 28 days post dose (Day 29), calculated by the linear trapezoidal method |
| AUC <sub>last</sub> | Area under the norbuprenorphine plasma concentration-time curve from time 0 (Day 1) to the last quantifiable concentration, calculated by the linear trapezoidal method |
| C <sub>max</sub> | Maximum observed norbuprenorphine plasma concentration |
| T <sub>max</sub> | Time to attain the maximum observed norbuprenorphine plasma concentration |
| C <sub>trough</sub> | Norbuprenorphine plasma concentration measured on Day 29 |

AUC<sub>last</sub> for both analytes, and AUC<sub>0-28 Days</sub> and  $C_{max}$  for norbuprenorphine will be analyzed using the same statistical model as described in Section 5.3.2.

# 5.6 Other Safety Analyses

#### 5.6.1 Extent of Exposure

Regarding the exposure to SUBOXONE in the Run-in Period, the following will be summarized for the Run-In safety and Safety Analyses Sets.

- The number of days of SUBOXONE use prior to randomization. The number of days will
  be calculated as the date of the last dose of SUBOXONE minus the date of the first dose
  of SUBOXONE plus 1.
- The total SUBOXONE dose and average daily SUBOXONE dose during the entire run-in period, calculated as the total cumulative dose divided by the number of days of use.
- The total SUBOXONE dose and average daily SUBOXONE dose between day -7 and day -1.

#### 5.6.2 Adverse Events

Treament Emergent Adverse Events (TEAEs) are defined as adverse events with a start time that is equal to or later than the initiation of the drug treatment or any event already present that worsens in either intensity or frequency following drug exposure.

TEAEs with start date-time after the date of the 1<sup>st</sup> SUBOXONE dose and before the date of SUBLOCADE injection will be reported for the run-in period, using run-in safety and Safety Analysis Set.

TEAEs with start date-time equal to or after SUBLOCADE injection will be reported for the post-injection period, using Safety Analysis Set, by actual injection site and overall.

TEAEs will be coded to system organ class (SOC) and preferred term (PT) using MedDRA. Incidence and incidence proportion of TEAE (number and percentage of participants reporting the TEAE at least once during the run-in period or the post-injection period) and TEAEs identified as injection site reactions (post-injection period only) will be summarised by SOC and PT. Separate summaries will be provided for the two periods for all TEAEs, TEAEs identified as injection site reactions (post-injection period only), Serious TEAEs, drug related TEAEs and TEAEs leading to discontinuation of study treatment (SUBOXONE or SUBLOCADE).

TEAEs will also be summarized by maximum severity and relatedness within SOC and PT. If an AE is reported more than once by a subject within a SOC and/or PT, the maximum reported level of severity/relatedness will be used at each level of summation in the severity/relationship summary tables. Missing severity and relatedness will be queried until resolution. If resolution is not possible, missing severity will be summarized as "severe" and missing relatedness will be summarized as "related."

#### 5.6.3 Additional safety assessments

#### 5.6.3.1 Laboratory Data

Except for the pregnancy test which is done both at screening and upon admission to the clinical site, all laboratory evaluations (Table 7) at screening will be summarized using both the Run-In safety and the Safety Analysis Set. Liver function tests will be summarized by time point, using Safety Analysis Set. In calculating summary statistics for numeric lab test values, any reported value that include qualifiers (ie, <,  $\le$ , >) will be summarized as the limit of quantification. E.g. > 9 will be summarized as 9.

Pregnancy test results will only be listed.

**Table 7. Laboratory Assessments** 

| Laboratory<br>Assessments | Parameters | |
|---|---|---|
| Haematology | Platelet count | |
| | Red blood cell (RBC) count | |
| | - | cular volume (MCV)<br>cular haemoglobin (MCH) |
| | White blood cell (WBC) count with differential: | <ul><li>Neutrophils</li><li>Lymphocytes</li><li>Monocytes</li><li>Eosinophils</li><li>Basophils</li></ul> |
| | Haemoglobin | |
| | Haematocrit | |
| Clinical Chemistry | Blood urea nitrogen (BUN) Potassium Creatinine Sodium Calcium | Bicarbonate Chloride Glucose (fasting or non-fasting) Creatine phosphokinase (CPK) |
| Liver Function Test | Albumin Lactate dehydrogenase (LDH) Total protein Aspartate aminotransferase (AST) Alanine aminotransferase (ALT) Alkaline phosphatase (ALP) Gamma glutamyl transferase (GGT) Total and direct bilirubin | |
| Pregnancy Testing | Highly sensitive urine human chorio test (as needed for women of childb | |
| Urine Drug Screen | Opioids Cocaine Fentanyl Oxycodone Opiates/Morphine Amphetamines Methadone Cannabinoids Barbiturates Benzodiazepines Methamphetamine Phencyclidine | |

| Other Laboratory | Serology (HIV-1 and -2 antibodies, hepatitis B surface antigen [HbsAg], |
|---|---|
| Tests | and hepatitis C virus antibody, PTT, and PT with INR) If a central |
| | laboratory is being utilised and protocol-required additional local |
| | laboratory assessments are needed, include the last bullet in the Other |
| | screening tests section of the table ([All study required laboratory): |
| Urinalysis | Specimen Appearance, Bilirubin, Color, Glucose, Ketone, Leucocyte |
| (Categorical) | Esterase, Nitrite, Occult Blood, Protein, Urobilinogen, Erythrocytes, |
| | Leukocytes |
| Urinalysis | pH, Specific Gravity. |
| (Continuous) | |

#### **5.6.3.2** Vital signs

Vital signs (systolic and diastolic blood pressure, pulse rate, respiratory rate) will be summarized by time point, using the Safety Analysis Set and Run-In Safety Set.

#### 5.6.3.3 ECG data

ECG interpretation (normal, abnormal but not clinically significant, abnormal and clinically significant) will be summarized by time point. Numeric 12-lead ECG parameters [heart rate, PR interval, QRS duration, QT interval, Fridericia's corrected QT interval (QTcF)] will also be summarized. All summaries will be based on the Safety Analysis Set and Run-In Safety Set.

#### 5.7 Other Analyses

#### 5.7.1 Major Protocol Deviations

Major protocol deviations will be identified and documented prior to database lock and will be summarized by category (eg, prohibited medication, out-of-window assessment), per the Protocol Deviation Plan for the study, for screened subjects. Deviations that occur in subjects who were randomized and not randomized will be summarized separately. All major protocol deviations will be listed.

#### 5.7.2 Demographic and Baseline Disease Characteristics

Demographic and other baseline characteristics will be summarized separately for the run-in safety set, safety set and PK Evaluable Set, if different. Parameters to be summarized will be age, sex, race, ethnicity, fertility status, and height/weight/body mass index, drug use history and route of administration.

# 5.7.3 Medical and Psychiatric History

Relevant medical history will be coded using MedDRA and will be summarized for the Run-In Safety population and safety population (PK population, if different).

#### 5.7.4 Urine Drug Screen Results

The number and percentage of participants with positive UDS will be summarized by time point, using the Run-In safety analysis set and Safety Analysis Set. The denominator of the percentage is the number of participants with available results for the individual drug. The opioids (overall) will include opiates/morphine, methadone, oxycodone, and fentanyl. If any of these are "Positive", then opioids (overall) will be defined as "Positive". If all non-missing test results are negative, then opioids (overall) will be defined as "Negative". Amphetamine and methamphetamine will be combined into one class as amphetamine/methamphetamine, using the similar definition for "Positive/Negative" as opioids (overall).

# 5.7.5 Prior and Concomitant Therapies and Medications

Therapies and medications will be collected from screening through EOS and will be coded using Anatomical Therapeutic Chemical (ATC) classification codes via the World Health Organization Drug Dictionary (WHO-DD). Prior and concomitant medications during run-in/post-injection period are defined in Appendix 8: Concomitant Medication Definition.

Prior and concomitant medications will be summarized using the run-in safety and safety populations. Concomitant medications during the run-in and post-injection periods will be summarized separately using the run-in safety and safety populations, respectively. The summary of incidence (number and percentage of subjects reporting the medication at least once) will be sorted alphabetically by therapeutic class (ATC level 3) and standardized medication name.

#### 5.7.6 Subgroup analyses

In order to understand the study site-to-site variation in injection technique and assessment of injection site reactions, injection site grading and injection site pain VAS summary tables will be repeated for each study site.

#### 5.8 Interim Analyses

Not applicable.

#### 6 SUPPORTING DOCUMENTATION

#### **6.1** Appendix 1: List of Abbreviations

**Table 8. List of Abbreviations** 

| Abbreviation | Definition |
|--------------|---------------------------------|
| AE | adverse event |
| ANOVA | Analysis of variance |
| ATC | Anatomic Therapeutic Chemical |
| AUC | area under the curve |
| BLQ | below the limit of quantitation |
| BP | blood pressure |

| Abbreviation | Definition |
|------------------|----------------------------------------------|
| BUP | buprenophine |
| CI | confidence interval |
| C <sub>max</sub> | maximum observed concentration |
| CMQ | customised MedDRA queries |
| CSR | clinical study report |
| ECG | electrocardiogram |
| ICF | Informed consent form |
| MedDRA | Medical Dictionary for Regulatory Activities |
| PK | pharmacokinetic(s) |
| PT | preferred term |
| QT | QT |
| QTcF | corrected QT (Fridericia method) |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SD | standard deviation |
| SOC | System Organ Class |
| TEAE | treatment-emergent adverse event |

# 6.2 Appendix 2: Changes to Protocol-Planned Analyses

Not applicable.

# 6.3 Appendix 3: Definition and Use of Visit Windows in Reporting

Regardless of any actual blood draw time deviations from the scheduled time, summary statistics by time point (for data tabulations and figures) will use the scheduled time point.

# 6.4 Appendix 4: Endpoint Derivations

#### 6.4.1 PK Parameters

Plasma PK parameters will be calculated by non-compartmental analysis using WinNonlin software for BUP and norbuprenorphine. Actual sampling times will be used in the calculations.

If quantifiable data are not available through 28 days ( $T_{last}$  <28 days), the following rules will be used to extrapolate AUC<sub>0-28 Days</sub> from AUC<sub>last</sub> via linear regression through the terminal log-linear segment of the plasma concentration-time curve:

- At least three quantifiable concentrations will be used in the regression
- C<sub>max</sub> or data prior to C<sub>max</sub> will not be included in the regression.
- The adjusted regression coefficient ( $R^2$  adj) should be  $\ge 0.80$ .

#### 6.4.2 Handling of BLQ and abberant plasma concentrations

Plasma concentrations that are below the lower limit of quantification (BLQ) will be treated as zero for the time point summary statistics and linear-scale plots of concentrations and excluded from semi-logarithmic-scale plots of concentrations.

For deriving BUP and norbuprenorphine PK parameters, all plasma concentrations that are BLQ prior to the peak plasma concentration ( $C_{max}$ ) will be set to zero. Post  $C_{max}$ , BLQ values will be handled as follows:

- Embedded BLQ values that are between two measurable concentrations will be set to missing
- Measurable concentrations between two BLQ values will be set to missing
- If two or more consecutive BLQ concentrations are followed by quantifiable concentrations, these quantified values will be set to missing
- If a BLQ concentration is followed by a quantifiable concentration, and the quantifiable concentration is then followed by two or more consecutive BLQ concentrations, the quantifiable concentration will be set to missing
- Terminal BLQ values following the last quantifiable time point will be set to missing
- No concentration estimates will be imputed for missing sample values.

# 6.4.3 Injection site Reactions Customised MedDRA Queries (CMQ)

The PTs used to categorize the injection site reactions are shown in **Table 9** below.

Table 9 CMQ List of Preferred Terms for Injection Site Reactions

| Preferred Term | Preferred Term |
|---|---|
| Immediate post-injection reaction | Injection site ulcer |
| Injection related reaction | Injection site urticaria |
| Injection site abscess | Injection site vesicles |
| Injection site cellulitis | Injection site warmth |
| Injection site infection | Injection site ischaemia |
| Injection site pustule | Injection site coldness |
| Injection site abscess sterile | Injection site discolouration |
| Injection site anaesthesia | Injection site photosensitivity reaction |
| Injection site atrophy | Injection site swelling |
| Injection site bruising | Injection site discomfort |
| Injection site cyst | Injection site calcification |
| Injection site dermatitis | Injection site movement impairment |
| Injection site erosion | Injection site lymphadenopathy |
| Injection site erythema | Injection site nodule |
| Injection site extravasation | Embolia cutis medicamentosa |
| Injection site fibrosis | Injection site scar |
| Injection site granuloma | Injection site discharge |
| Injection site haematoma | Injection site pallor |
| Injection site haemorrhage | Injection site papule |
| Injection site hypersensitivity | Injection site injury |
| Injection site hypertrophy | Injection site scab |
| Injection site induration | Injection site eczema |

| Injection site inflammation | Injection site streaking |
|-----------------------------|-------------------------------|
| Injection site irritation | Injection site dryness |
| Injection site mass | Injection site laceration |
| Injection site necrosis | Injection site macule |
| Injection site nerve damage | Injection site vasculitis |
| Injection site oedema | Injection site exfoliation |
| Injection site pain | Injection site dysaesthesia |
| Injection site paraesthesia | Injection site plaque |
| Injection site phlebitis | Injection site hyperaesthesia |
| Injection site pruritus | Injection site hypoaesthesia |
| Injection site rash | Injection site hypertrichosis |
| Injection site reaction | Injection site thrombosis |

# 6.5 Appendix 5: Methods to Manage Missing Data

#### 6.5.1 Adverse event data

# **Missing AE Severity**

In the unlikely event that resolution is not possible, missing severity will be imputed as "severe" in summaries.

#### Missing AE Relationship to Study Drug

In the unlikely event that resolution is not possible, missing relationship will be imputed as "related" in summaries.

#### **Missing Date Information for Adverse Events**

- Missing day and month
  - If the year is the same as the year of the date of the first dose of investigational product, then the day and month of the date of the first dose of investigational product will be assigned to the missing fields.
  - If the year is before the year of the date of the first dose of investigational product, then December 31 will be assigned to the missing fields.
  - If the year is after the year of the date of the first dose of investigational product, then January 1 will be assigned to the missing fields.
- Missing month only
  - The day will be treated as missing and both month and day will be replaced according to the above procedure.
- Missing day only

- If the month and year are the same as the month and year of the date of the first dose of investigational product, then the day of the first dose of investigational product will be assigned to the missing day.
- If either the year is before the year of the date of the first dose of investigational product or if both years are the same but the month is before the month of the date of the first dose of investigational product, then the last day of the month will be assigned to the missing day.
- If either the year is after the year of the date of the first dose of investigational product or if both years are the same but the month is after the month of the date of the first dose of investigational product, then the first day of the month will be assigned to the missing day.
- If the stop date is after the date of the first dose of investigational product, the date of the first dose of investigational product will be assigned to the missing start date.
- If the stop date is before the date of the first dose of investigational product, the stop date will be assigned to the missing start date.

#### 6.5.2 Missing Date Information for Concomitant Medications

- Missing day and month
  - If the year of the incomplete start date is the same as the year of the date of the first dose of investigational product, then the day and month of the date of the first dose will be assigned to the missing fields.
  - If the year of the incomplete start date is before the year of the date of the first dose of investigational product, then December 31 will be assigned to the missing fields.
  - o If the year of the incomplete start date is after the year of the date of the first dose of investigational product, then January 1 will be assigned to the missing fields.

#### Missing month only

 The day will be treated as missing and both month and day will be replaced according to the above procedure.

# Missing day only

- If the month and year of the incomplete start date are the same as the month and year of the date of the first dose of investigational product, then the day of the first dose will be assigned to the missing day.
- If either the year is before the year of the date of the first dose of investigational product or if both years are the same but the month is before the month of the date of the first dose of investigational product, then the last day of the month will be assigned to the missing day.
- If either the year is after the year of the date of the first dose of investigational product or if both years are the same but the month is after the month of the date of the first dose of investigational product, then the first day of the month will be assigned to the missing day.

#### Incomplete Stop Date

 For deriving concomitant medication flag, the following rules will be applied to impute the missing numerical fields. If the date of the last dose of investigational product is missing, impute it as descripted in Section 17.4. If the imputed stop date is before the start date (imputed or non-imputed start date), then the imputed stop date will be equal to the start date.

#### Missing day and month

- If the year of the incomplete stop date is the same as the year of the date of the last dose of investigational product, then the day and month of the date of the last dose will be assigned to the missing fields.
- If the year of the incomplete stop date is before the year of the date of the last dose of investigational product, then December 31 will be assigned to the missing fields.
- If the year of the incomplete stop date is after the year of the date of the last dose
  of investigational product, then January 1 will be assigned to the missing fields.

#### Missing month only

 The day will be treated as missing and both month and day will be replaced according to the above procedure.

# Missing day only

- If the month and year of the incomplete stop date are the same as the month and year of the date of the last dose of investigational product, then the day of the last dose will be assigned to the missing day.
- If either the year is before the year of the date of the last dose of investigational product or if both years are the same but the month is before the month of the date of the last dose of investigational product, then the last day of the month will be assigned to the missing day.
- If either the year is after the year of the date of the last dose of investigational product or if both years are the same but the month is after the month of the date of the last dose of investigational product, then the first day of the month will be assigned to the missing day.

#### 6.6 Appendix 6: Methods to Manage Character Values of Clinical Laboratory Parameters

Reported values of clinical laboratory parameters that include qualifiers (ie, <,  $\le$ , >,  $\ge$ ) will be listed as reported but will be summarized without the qualifier.

# 6.7 Appendix 7: Data Set Descriptions

Trial data sets will consist of CRF exports and external data files. External files may be used for PK parameters, protocol deviations and data from the central laboratory, for example.

#### 6.8 Appendix 8: Concomitant Medication Definition

The definition of prior and concomitant medications is illustrated below. Two timing flags will be derived based on the tables below.

Table 10 Definition of Prior and Concomitant Medications for Run-In Period

| End Date of Non-Study | Start Date of Non-Study Medication | | |
|---|---|---|---|
| Medication | Missing | < Start date of | ≥ Start date of SUBOXONE and ≤ |
| Wedication | | SUBOXONE | end date of SUBOXONE |
| Missing (includes flagged as "Ongoing") | Prior<br>Concomitant (Run-In) | Prior<br>Concomitant (Run-In) | Concomitant (Run-In) |
| < Start date of SUBOXONE | Prior | Prior | Data Error |
| ≥ Start date of SUBOXONE<br>and ≤ end date of<br>SUBOXONE | Prior<br>Concomitant (Run-In) | Prior<br>Concomitant (Run-In) | Concomitant (Run-In) |

If a medication's end date is on or after the date of SUBLOCADE injection, then it will be classified as concomitant Post-Injection as shown in Table 11.

**Table 11 Definition of Concomitant Medications for Post Injection Period** 

| End Date of Non-Study | Start Date of Non-Study Medication | | |
|---|---|---|---|
| Medication | Missing | < SUBLOCADE injection date | ≥ SUBLOCADE injection date |
| Missing (includes flagged as "Ongoing") | Concomitant (Post-<br>Injection) | Concomitant (Post-Injection) | Concomitant (Post-Injection) |
| ≥ SUBLOCADE injection date | Concomitant (Post-<br>Injection) | Concomitant (Post-Injection) | Concomitant (Post-Injection) |

Prior medications will be defined using the first table only. A medication is considered concomitant if it is concomitant either during run-in period or during post-injection period.

# 7 REFERENCES

- 1. Phoenix™ WinNonlin® (Version 8.3.4.295 or higher, Certara, LP.)
- 2. Certara Integral (Version 22.10.1, Certara, USA, Inc.)
- 3. SAS Institute Inc., Cary, NC, 27513, USA